CLINICAL TRIAL: NCT06638554
Title: Integrating Telehealth to Advance Lung Cancer Screening
Acronym: ITALCS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Katharine Rendle, Associate Professor, Abramson Cancer Center at Penn Medicine
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Health Services Research
Other Study IDs: UPCC 04524; P50CA271338 (NIH); 850376 (Other: Penn IRB)
Record Dates: First submitted 2024-10-09; First posted 2024-10-15 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Early Detection of Cancer; Telemedicine; Decision Making

STUDY DESIGN:
Intervention Model Description: This study uses a sequential randomization design in which all eligible participants will be randomized into one of two interventions at Stage 1 and then participants that do not respond to Stage 1 interventions will be randomized to receive Stage 2 interventions
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Active Choice (Stage 1) + Low Touch (Stage 2) (Experimental): Participants in this arm will be offered the option via outreach letter to complete an SDM visit via telehealth or in-person (Stage 1) and if individuals do not schedule an SDM visit within 30 days (non-responders), they will receive asynchronous text messages alone (Stage 2)
  Interventions: Behavioral: Active Choice; Behavioral: Low Touch Strategy
- Active Choice (Stage 1) + High Touch (Stage 2) (Experimental): Participants in this arm will be offered the option via outreach letter to complete an SDM visit via telehealth or in-person (Stage 1) and if individuals do not schedule an SDM visit within 30 days (non-responders), they will receive asynchronous text messages in combination with synchronous digital care coordination (Stage 2).
  Interventions: Behavioral: Active Choice; Behavioral: High Touch Strategy
- Telehealth Only (Stage 1) + Low Touch (Stage 2) (Experimental): Participants in this arm will be offered the option via outreach letter to complete an SDM visit via telehealth only (Stage 1) and if individuals do not schedule an SDM visit within 30 days (non-responders), they will receive asynchronous text messages alone (Stage 2).
  Interventions: Behavioral: Telehealth Only; Behavioral: Low Touch Strategy
- Telehealth Only (Stage 1) + High Touch (Stage 2) (Experimental): Participants in this arm will be offered the option via outreach letter to complete an SDM visit via telehealth only (Stage 1) and if individuals do not schedule an SDM visit within 30 days (non-responders), they will receive asynchronous text messages in combination with synchronous digital care coordination (Stage 2).
  Interventions: Behavioral: Telehealth Only; Behavioral: High Touch Strategy

INTERVENTIONS:
Behavioral: Active Choice — The participant will be send a letter inviting them to complete a SDM visit either in-person or via telehealth.
  Arms: Active Choice (Stage 1) + High Touch (Stage 2); Active Choice (Stage 1) + Low Touch (Stage 2)
Behavioral: Telehealth Only — The participant will be send a letter inviting them to complete a SDM visit via telehealth only.
  Arms: Telehealth Only (Stage 1) + High Touch (Stage 2); Telehealth Only (Stage 1) + Low Touch (Stage 2)
Behavioral: Low Touch Strategy — Patient will be sent asynchronous text messaging reminders encouraging SDM for LCS using framed messaging.
  Arms: Active Choice (Stage 1) + Low Touch (Stage 2); Telehealth Only (Stage 1) + Low Touch (Stage 2)
Behavioral: High Touch Strategy — Patient will be sent asynchronous text messaging reminders encouraging SDM for LCS using framed messaging in combination with synchronous telephone-based digital care coordination.
  Arms: Active Choice (Stage 1) + High Touch (Stage 2); Telehealth Only (Stage 1) + High Touch (Stage 2)

SUMMARY:
The goal of this pragmatic trial is to learn if telehealth strategies can increase shared decision-making (SDM) for lung cancer screening (LCS). It will also learn about the equity of these strategies by conducting non-inferiority analysis by race and sex. The main questions it aims to answer are:

1. Does patient outreach using synchronous and asynchronous telehealth strategies increase completion of SDM visits for LCS?
2. Is the effectiveness of these telehealth strategies similar by race and sex?

The study uses a Sequential Multiple Assignment Randomized Trial (SMART) design and includes two stages of interventions. The first stage of intervention includes direct patient outreach with an invitation to schedule either a 1) telehealth SDM visit or 2) telehealth or in-person SDM visit. Participants that do not respond to the first stage interventions receive a text message reminder encouraging SDM visit completion with or without digital care coordination.

DETAILED DESCRIPTION:
Annual lung cancer screening using low-dose computed tomography (LDCT) is associated with decreased lung cancer mortality but also with harms. As such, it is recommended, and required for reimbursement, that patients complete an shared decision-making visit (SDM) prior to screening to discuss potential risks and benefits in the context of patient values. Despite guidelines recommending screening and national insurance coverage of LDCT, uptake of SDM visits and subsequent LDCT is remarkably low. We aim to address these gaps by comparing the effectiveness of synchronous and asynchronous telehealth strategies on SDM visits and subsequent LDCT in a pragmatic trial using a Sequential Multiple Assignment Randomized Trial (SMART) design. The specific first stage strategies to be tested are: a) Active Choice Outreach (invitation to schedule a telehealth or in-person SDM visit) vs b) Telehealth Only Outreach (invitation to schedule a telehealth SDM visit). The specific second stage strategies (delivered only if participants do not respond to first stage interventions) are a) text message reminders encouraging SDM visit completion (low-touch) alone or b) in combination with phone-based digital care coordination (high-touch). We will also assess non-inferiority of strategies by race and sex to assess equity of effectiveness.

ELIGIBILITY:
Inclusion criteria:

Participants will be eligible if:

1. are aged 50 to 80
2. have a history of tobacco use indicated by either: Documented 20 pack-year or greater smoking history in their electronic health record (EHR); OR Self-report via structured survey
3. currently smoke or formerly smoked cigarettes
4. have no documented history of lung cancer
5. have no documented history of lung cancer screening in the 24 months prior to study enrollment
6. have completed at least one primary care visit at Penn Medicine in the 3 years prior to study enrollment.

Exclusion criteria:

Participants who do not meet inclusion criteria will not be eligible.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6000 (Estimated)
Dates: Start 2024-07-09 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Shared decision making (SDM) for lung cancer screening (LCS) | 90 days after randomization
  Completion of an SDM visit (in person or telehealth) defined as any completed encounter that has documented SDM for LCS as indicated by 1) procedure code (G0296 or equivalent), or documentation of SDM conversation related to LCS in associated progress notes.

SECONDARY OUTCOMES:
Low-dose computed tomography (LDCT) | 6 months after randomization
  Completion of LDCT within 6 months of randomization date among individuals who complete SDM and are determined to be eligible for LCS.

OTHER OUTCOMES:
Fidelity to Shared Decision-Making | Up to 90 days after randomization
  Completion of key components of SDM for LCS including:
  1. discussion of risks & benefits of LCS
  2. use of decision aid
  3. elicitation of patient preferences
  4. tobacco cessation support
Fidelity to Digital Care Coordination | Up to 90 days after randomization
  Completion of key components of digital care coordination including assessing digital needs and readiness, providing technological support, answering questions about security or safety, and helping to coordinate telehealth appointments.
Lung cancer diagnoses | 12 months after randomization
  Number of people diagnosed with lung cancer after randomization.
Reach: Text Message Delivery | Up to 90 days after randomization
  The number of participants who are successfully delivered text messages divided by those who are sent text messages in Stage 2.
Reach: Digital Care Coordination | Up to 90 days after randomization
  The number of participants who complete a digital care coordination visit divided by those contacted by the Digital Care Coordinator in Stage 2.
Reach: Scheduling | Up to 90 days after randomization
  The number of participants who schedule an SDM visit divided by those who are sent initial outreach.
Timeliness | Up to 12 months after randomization
  The number of days between randomization and SDM completion among subjects who complete SDM for LCS.

CONTACTS AND LOCATIONS:
Overall Officials: Katharine Rendle, PhD, Principal Investigator — Abramson Cancer Center
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No